CLINICAL TRIAL: NCT02360917
Title: Emerging From the Haze™-A Multi-center, Randomized Controlled Trial to Measure Impact of a Multi-dimensional Psycho-educational Program on Subjective Cognitive Complaints After Breast Cancer Treatment Using Virtual Technology
Brief Title: Emerging From the Haze™- Measuring the Impact of a Psycho-education Program on Perceived Cognition After Breast Cancer Treatment
Acronym: Haze
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: University of Kansas (Other); University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Arash Asher, MD, Director, Cancer Survivorship and Rehabilitation Samuel Oschin Comprehensive Cancer Institute Cedars-Sinai Medical Center, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IIT 2014-01
Record Dates: First submitted 2015-02-06; First posted 2015-02-11 (Estimated); Last update posted 2018-11-01 (Actual); Status verified 2018-10

CONDITIONS: Cognition; Cancer
Keywords: Cognitive Dysfunction; Cancer Survivorship
MeSH Terms: conditions — Neoplasms; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Participants in the intervention group will undergo 6 weeks of psycho-educational classes provided in a live setting at Cedars Sinai and a web based setting at The University of Kansas. Each class will focus on a different realm of coping with chemo-brain.
  Interventions: Other: Emerging from the Haze
- Waitlist (Other): Participants assigned to the control group will be placed on a wait list for the Haze program. While they are waiting for admittance to the program, they will receive the same surveys as the participants who are taking the Haze class. Additionally, participants assigned to the control group will receive the surveys again when taking the class in order to allow comparison of the effects of the program on the control group. Participants assigned to the wait list will be enrolled in the following Haze series.
  Interventions: Other: Emerging from the Haze

INTERVENTIONS:
Other: Emerging from the Haze — A 6 week psycho-educational class

SUMMARY:
At Cedars-Sinai Medical Center, we have developed a novel curriculum for a 6-week psycho-educationally-based, cognitive behavioral program to help patients with subjective cognitive complaints after cancer treatment, titled Emerging from the Haze™ (Haze). Each series meets once a week for 2 hours for 6 weeks. The leading neuropsychologist covers material such as guided relaxation, behavioral strategies for automatic/negative thoughts, compensatory strategies for attention and memory, executive functioning, pacing, and balance. Each Haze series will be electronically delivered in a live format to our satellite site, The University of Kansas.

ELIGIBILITY:
Inclusion Criteria:

* Completed treatment for stage 1-3 breast cancer at least two months but not more than 24 months prior to enrollment.
* Having received chemotherapy with or without radiation therapy
* Female, Age ≥18 years.
* FACT-Cog score less than 59 on the Perceived Cognitive Impairment subscale
* Eligible after 2 months of completing all their active cancer treatment with the exception of long-term hormonal treatments or trastuzumab.
* Subjective complaint of cognitive concerns at time of enrollment
* Must be able to understand and communicate proficiently in English
* Ability to understand and the willingness to sign a written informed consent.
* Agree to complete study surveys

Exclusion Criteria:

* Patients who have significant personality disorders or unstable psychiatric disorders (including active major depression, substance abuse, psychosis or bipolar disorder) as assessed by the interviewing clinician
* Patients with known brain metastases, history of brain metastases or radiation to the brain.
* Patients with a history of stroke or other pre-existing neurological condition that may contribute to cognitive dysfunction.
* Non-English speakers
* Receiving treatment for another malignancy other than breast cancer
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, chronic anemia, uncontrolled hypothyroidism, symptomatic congestive heart failure, unstable angina pectoris, uncontrolled cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2015-07-06 (Actual); Primary Completion 2018-03-17 (Actual); Study Completion 2018-05-23 (Actual)

PRIMARY OUTCOMES:
quantify the impact of Emerging from the Haze on breast cancer survivors' self-report of cognitive changes, based on change of the FACT-Cog- perceived cognitive impairment score from baseline to the end of the Haze series compared to the control group. | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Myers, PhD, RN AOCNSP, Principal Investigator — University of Kansas; Arash Asher, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States